CLINICAL TRIAL: NCT05391087
Title: Comparison of Arterial Blood Pressure and Cardiac Index-based Hemodynamic Management on Postoperative Myocardial Injury in Patients Undergoing Hepatopancreatic Surgery: a Randomized Clinical Trial
Brief Title: Comparison Arterial Blood Pressure and Cardiac Index-based Hemodynamic Management on Postoperative Myocardial Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Saglik Bilimleri University (Other)
Responsible Party: Principal Investigator, Taner Abdullah, Medical Doctor, Istanbul Saglik Bilimleri University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2021.12.271
Record Dates: First submitted 2022-05-20; First posted 2022-05-25 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-07

CONDITIONS: Myocardial Injury; Perioperative/Postoperative Complications
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mean Arterial Pressure (MAP) Group (Active Comparator): Target MAP: Baseline MAP +/- 20% and MAP>65mmHg Baseline MAP: MAP average in the ward at rest the day before surgery Low MAP intervention If PPV>14, apply 500ml crystalloid If PPV>9 and any additional finding regarding hypovolemia, apply 500ml crystalloid If PPV<10, start/titrate noradrenaline infusion
  Interventions: Other: Mean arterial pressure based management
- Cardiac Index (CI) Group (Active Comparator): CI: Baseline CI +/- 20% and CI > 2.2 L/m2/min Baseline CI: CI calculated by MostCare monitor before the anesthesia induction starts Low CI intervention If PPV>9, apply mini fluid challenge (MFC). If MFC is positive, apply 500ml crystalloid.
  If MFC is negative, evaluate MAP. If MAP is elevated start/titrate remifentanil. If MAP is not elevated start/titrate dopamine/dobutamine in accordance with systemic vascular resistance index (SVRI)
  Interventions: Other: Cardiac index based management

INTERVENTIONS:
Other: Mean arterial pressure based management — Mean arterial pressure group: Low MAP will be intervened in accordance with the protocol as described in the arm
  Arms: Mean Arterial Pressure (MAP) Group
Other: Cardiac index based management — Cardiac index group: Low CI will be intervened in accordance with the protocol as described in the arm. Additionally, if MAP is lower than target MAP along with a normal CI, this will be intervened with noradrenalin infusion/titration
  Arms: Cardiac Index (CI) Group

SUMMARY:
The primary aim of this study is to compare mean arterial pressure (MAP) and cardiac index (CI) based intraoperative hemodynamic management in terms of postoperative high sensitive troponin elevation.

The hypothesis of the study is that there will be at least 5ng/L difference between the two groups in terms of troponin elevation occurring in the postoperative period. When power analysis was performed with this primary output, it was calculated that while alpha was 0.05 beta 0.2, 42 patients in each group, a total of 84 patients were required.

DETAILED DESCRIPTION:
Fluid therapy will be started as 2-4 ml/kg/h, according to the clinician's decision for the patient. Afterwards, patients will be managed hemodynamically with one of the MAP and CI algorithms.

Targeted fluid therapy will be administered in accordance with the following definitions of normal and algorithms for both groups.

Normal definitions:

MAP: Baseline MAP +/- 20% and MAP>65mmHg Baseline MAP: MAP average in the ward at rest the day before surgery

CI: Baseline CI +/- 20% and CI > 2.2 L/m2/min Baseline CI: CI calculated by MostCare monitor before the anesthesia induction starts

Low MAP intervention If PPV>14, apply 500ml crystalloid If PPV>9 and any additional finding regarding hypovolemia, apply 500ml crystalloid If PPV<10, start/titrate noradrenaline infusion

Low CI intervention If PPV>9, apply mini fluid challenge (MFC). If MFC is positive, apply 500ml crystalloid.

If MFC is negative, evaluate MAP. If MAP is elevated start/titrate remifentanil. If MAP is not elevated start/titrate dopamine/dobutamine in accordance with SVRI

ELIGIBILITY:
Inclusion Criteria:

1. Patients who will undergo pancreatic-hepatic surgery
2. Patients over 65 years of age or patients over 45 years of age and with at least one of the following comorbidities:

coronary artery disease, Congestive heart failure, moderate to severe heart valve disease, peripheral artery disease Moderate to Severe Pulmonary hypertension, cerebrovascular accident older than 1 month, History of pulmonary embolism more than 1 month old, Diabetes Mellitus, Hypertension

Exclusion Criteria:

1. Presence of atrial fibrillation, sepsis, pulmonary embolism
2. Presence of pulmonary embolism, acute coronary syndrome and cerebrovascular accident in the last month
3. Static respiratory system compliance < 35ml/cmH2O
4. Patients with preoperative high sensitive Troponin T value >65ng/liter
5. glomerular filtration rate < 60 ml/min

Exclusion criteria during the protocol:

1. Newly developed arrhythmia, embolism, sepsis,
2. Cancellation of planned surgery
3. Postoperative hepatic failure defined as INR>2

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-03-28 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Postoperative high sensitive troponin change | three days
  difference between the mean high sensitive troponin elevation between the groups will be evaluated. high sensitive troponin T will be measured one day before the surgery, and daily after the surgery for three days

SECONDARY OUTCOMES:
postoperative myocardial injury incidence | three days
  high-sensitivity troponin T elevation by at least 5 ng/L from the preoperative concentration to at least 20 ng/L
90-days mortality | 90 days
  comparison of mortality frequency on the 90th day of the surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Başakşehir Çam and Sakura City Hospital, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Derived] Abdullah T, Gokduman HC, Eniste IA, Kudas I, Ali A, Kinaci E, Ozden I, Gumus Ozcan F. Mean arterial pressure versus cardiac index for haemodynamic management and myocardial injury after hepatopancreatic surgery: A randomised controlled trial. Eur J Anaesthesiol. 2024 Nov 1;41(11):831-840. doi: 10.1097/EJA.0000000000002059. Epub 2024 Sep 12. PMID 39262319